CLINICAL TRIAL: NCT06644469
Title: Effects of Whole-Body Vibration on Bone Mineral Density, Hand Grip Strength, and Vitamin D Levels in Middle-Aged Men: a Preliminary Clinical Trial
Brief Title: Whole Body Vibration in Middle Aged Men
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jouf University (Other)
Responsible Party: Principal Investigator, Fahad Alanazi, Assistant professor, Jouf University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JoufU
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Bone Density; Muscle Weakness
Keywords: Pilot Study; Bone Density; Vibration Therapy; Vitamin D; Muscle Strength
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The participants will be unaware of whether they are receiving vibration therapy, and the individual performing the assessment will be different from the one administering the treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group with placebo vibration therapy (Placebo Comparator): Participants will perform the same activities as the experimental group, but with a vertical displacement of 0.22 mm, deemed therapeutically insufficient.
  Interventions: Device: Placebo Dynatronics VF5 Model vibration platform
- Experimental Group (Experimental): Participants will undergo an 8-week WBV therapy program using a Dynatronics VF5 Model vibration platform. Each session will last 4 minutes, with vibration frequencies progressively increased from 25 Hz to 40 Hz without rest intervals.
  Interventions: Device: Dynatronics VF5 Model vibration platform

INTERVENTIONS:
Device: Dynatronics VF5 Model vibration platform — The Dynatronics VF5 Model vibration platform is a specialized therapeutic device designed for rehabilitation and wellness applications. Utilizing advanced vibration technology, it provides whole-body vibration therapy that can enhance muscle strength, improve flexibility, and promote overall physical well-being. The platform features adjustable frequency and amplitude settings, allowing customization based on individual needs. Its user-friendly interface and robust, durable design make it suitable for both clinical and mobile therapy settings. Additionally, the compact and portable nature of the VF5 facilitates easy storage and transport, while safety features such as non-slip surfaces ensure user protection.
  Arms: Experimental Group
Device: Placebo Dynatronics VF5 Model vibration platform — Placebo intensity with vertical vibration of 0.2 mm
  Arms: Control Group with placebo vibration therapy

SUMMARY:
This study aims of this clinical trial is to evaluate the effect of an 8-week Whole Body Vibration (WBV) intervention on Bone Mineral Density (BMD), hand grip strength, and vitamin D levels in middle-aged men. Findings from this study will contribute to understanding whether WBV is a viable alternative to conventional exercise, especially for those with limitations in physical activity.

Study Objectives:

• Primary Objective: To assess the effectiveness of an 8-week WBV intervention in improving BMD, hand grip strength, and vitamin D levels compared to a placebo intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male participants aged 50 years or older
* Participants with physical activity or exercise program involvement
* Participants with no history of serious medical conditions such as tumors, fractures, epilepsy, cardiac disease, or stroke within the past year.
* Participants must be non-smokers and not receiving hormone or calcium supplement therapy

Exclusion Criteria:

* Participants unable to stand on the WBV platform
* Participants with conditions contraindicating vibration therapy
* Participants participating in other clinical trials

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Bone Density | 8 weeks
  Changes in BMD (measured by DXA scanner),
Grip Strength | 8 weeks
  hand grip strength (measured by a hand-held dynamometer)
Vitamin D | 8 weeks
  Vitamin D levels (measured by high-performance liquid chromatography).

CONTACTS AND LOCATIONS:
Overall Officials: Fahad Alanazi, PhD, Principal Investigator — Jouf University
Locations (1):
- prince Mutaib bin Abdulaziz hospital, Sakakah, Aljouf, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol